CLINICAL TRIAL: NCT07375927
Title: A Randomized Controlled Study Evaluating the Effect of Postoperative Kinesio Taping on Pain and Functional Recovery Following Arthroscopic Rotator Cuff Repair
Brief Title: Effect of Kinesio Taping After Rotator Cuff Surgery
Acronym: RCR-KT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olcay Yavuz (Other)
Collaborators: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Olcay Yavuz, Medical Doctor, Orthopedic Surgery Resident, Fatih Sultan Mehmet Training and Research Hospital
Organization: Fatih Sultan Mehmet Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCR-KT-2026
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tears; Shoulder Pain; Post Operative Pain
Keywords: Rotator Cuff Tears; Kinesio Taping; Arthroscopic Rotator Cuff Repair; Postoperative Rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to either a kinesio taping group or a control group.
Who Masked: Outcomes Assessor
Masking Description: The investigator responsible for postoperative clinical assessments is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping Group (Experimental): Participants in this group will receive standard postoperative rehabilitation following arthroscopic rotator cuff repair, in addition to kinesio taping applied for three weeks during the postoperative period.
  Interventions: Other: Kinesio Taping; Other: Standard Postoperative Rehabilitation
- Control Group (Active Comparator): Participants in this group will receive standard postoperative rehabilitation alone following arthroscopic rotator cuff repair, without the application of kinesio taping.
  Interventions: Other: Standard Postoperative Rehabilitation

INTERVENTIONS:
Other: Kinesio Taping — Application of kinesio taping to the operated shoulder during the postoperative period as an adjunct to standard rehabilitation.
  Arms: Kinesio Taping Group
Other: Standard Postoperative Rehabilitation — Standard postoperative rehabilitation program following arthroscopic rotator cuff repair.

SUMMARY:
The aim of this study is to evaluate whether postoperative kinesio taping provides additional benefits in pain reduction and functional recovery in patients who have undergone arthroscopic rotator cuff repair.

Patients diagnosed with rotator cuff tear who have undergone surgical treatment will be randomly assigned into two groups. One group will receive standard postoperative rehabilitation together with kinesio taping applied for three weeks, while the control group will receive standard postoperative rehabilitation alone.

Pain levels and shoulder function will be assessed during postoperative follow-up using commonly accepted clinical evaluation scales. The findings of this study are expected to contribute to a better understanding of the role of kinesio taping in the recovery process after rotator cuff surgery.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of postoperative kinesio taping on pain levels and functional recovery in patients who have undergone arthroscopic rotator cuff repair.

Patients aged between 18 and 70 years with clinical suspicion of rotator cuff tear on physical examination and a diagnosis established by magnetic resonance imaging, with the tear confirmed intraoperatively, will be included in the study.

After providing written informed consent, eligible patients will be randomly assigned into two groups in a 1:1 ratio using a computer-generated randomization list.

The intervention group will receive standard postoperative rehabilitation combined with kinesio taping applied for three weeks following surgery. The control group will receive standard postoperative rehabilitation alone.

The study is designed as a single-blinded randomized controlled trial. The investigator responsible for postoperative clinical assessments will be blinded to group allocation in order to minimize evaluation bias.

Pain intensity and functional outcomes will be assessed during postoperative follow-up using validated clinical outcome measures, including the Visual Analog Scale (VAS), the Shoulder Pain and Disability Index (SPADI), and the UCLA shoulder score. Shoulder range of motion will also be recorded.

Patients will be evaluated at postoperative day 1, month 1, and month 3. Clinical outcomes will be compared between the two groups, as well as within each group over time, to assess the recovery process after surgery.

The results of this study are expected to provide further insight into the potential role of kinesio taping as an adjunctive method in postoperative rehabilitation following arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 70 years
* Patients with clinical suspicion of rotator cuff tear on physical examination and a diagnosis established by magnetic resonance imaging, with intraoperative confirmation
* Patients with at least two positive impingement tests on physical examination (Jobe, Hawkins-Kennedy, Neer)
* Patients without a diagnosed psychiatric disorder
* Patients without a history or current diagnosis of cervical pathology
* Patients with a Visual Analog Scale (VAS) score of 3 or higher for at least 3 months prior to surgery
* Patients able to participate regularly in postoperative follow-up for a period of one year
* Patients who agree to participate voluntarily and provide written informed consent

Exclusion Criteria:

* History of shoulder dislocation
* History of fracture involving the shoulder or surrounding structures
* Inability to comply with postoperative treatment or attend regular follow-up visits
* Known skin hypersensitivity or allergy to kinesio taping
* Known rheumatologic or neurological disease
* History of previous shoulder or peri-shoulder surgery
* Presence of cervical disc pathology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analog Scale, VAS) | Postoperative day 1, month 1, and month 3.
  Pain intensity will be assessed using the Visual Analog Scale (VAS), where higher scores indicate greater pain.

SECONDARY OUTCOMES:
Shoulder Function (SPADI Score) | Postoperative day 1, month 1, and month 3.
  Shoulder function will be evaluated using the Shoulder Pain and Disability Index (SPADI), with higher scores indicating greater pain and disability.
Shoulder Function (UCLA Shoulder Score) | Postoperative day 1, month 1, and month 3.
  Shoulder function will be assessed using the UCLA shoulder score during postoperative follow-up.
Shoulder Range of Motion | Postoperative day 1, month 1, and month 3.
  Active shoulder range of motion will be measured during postoperative follow-up.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared other researchers.